CLINICAL TRIAL: NCT00706953
Title: A Phase II Single Arm Study of VELCADE and DOXIL (PLD) in Patients With Relapsed Multiple Myeloma Previously Treated With VELCADE
Brief Title: A Study of Bortezomib and Pegylated Liposomal Doxorubicin in Patients With Relapsed Multiple Myeloma Previously Treated With Bortezomib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015091; DOXILMMY2009
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: pegylated liposomal doxorubicin; VELCADE; DOXIL; relapsed; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Active Comparator)
  Interventions: Drug: bortezomib; pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: bortezomib; pegylated liposomal doxorubicin — 1.3 mg/m2 IV bolus on Days 1,4,8,11 of each 21-day cycle; 30 mg/m2 IV infusion on Day 4 of each 21 day cycle

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using pegylated liposomal doxorubicin and bortezomib in the treatment of patients with relapsed multiple myeloma who had been previously treated with bortezomib. Multiple myeloma is a cancer that begins in plasma cells, a type of white blood cell. These cells are part of the immune system, which helps protect the body from germs and other harmful substances. In time, myeloma cells collect in the bone marrow and in the solid parts of bone. Multiple myeloma treatment may include stem cell transplantation, however, not all patients with multiple myeloma are candidates for stem cell transplantation and many patients who receive transplants relapse. As a result, additional first and later-line therapeutic options are needed for patients who are not candidates for transplantation, or whose disease relapses after transplantation or other therapies. Pegylated liposomal doxorubicin in combination with bortezomib is approved for the treatment of patients with multiple myeloma who have not previously received bortezomib and have received at least one prior therapy. The combined use of pegylated liposomal doxorubicin and bortezomib in this study is designed to evaluate the overall response rate and safety in patients with multiple myeloma who have been previously treated with bortezomib.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the overall response rate to DOXIL/VELCADE treatment in patients with relapsed multiple myeloma previously treated with VELCADE. Overall response rate is defined as the proportion of patients achieving either a complete response (CR) or partial response (PR) to treatment according to the European Group for Blood and Marrow Transplantation (EBMT) criteria. This is a single arm (all patients will receive the same drug combination and dose), multi-center (many study sites), open label (the patient and the physician know the drug treatment being received) of approximately 60 patients with multiple myeloma whose disease has progressed after initial response to VELCADE-based therapy. During each 21-day treatment cycle, patients will receive VELCADE by intravenous bolus on 4 designated days, and DOXIL by intravenous infusion on one designated day. Treatment will continue until disease progression, or the occurrence of unacceptable treatment-related toxicity or up to a total of 8 cycles of therapy. Drug doses may be delayed or dropped as needed to allow for platelet transfusions or other treatment requirements. Patients responding to treatment at study end may be evaluated for continued treatment for as long as treatment can be tolerated and they continue to respond. After discontinuation of all study drugs, patients who have not had disease progression will be followed for 6 months after receiving the last dose of study drug. The primary endpoint is overall response rate as defined by the proportion of patients achieving either a complete response or a partial response. Response will be assessed at each cycle. Safety will be monitored throughout the study by physical examination, clinical laboratory testing, and the incidence and severity of reported adverse events. Overall safety will be summarized at study-end.

During each 21-day treatment cycle, patients will receive bortezomib 1.3 mg/m2 by intravenous bolus on Days 1, 4, 8 and 11 and pegylated liposomal doxorubicin 30 mg/m2 by intravenous infusion on Day 4.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Myeloma
* Received prior courses of bortezomib (VELCADE)-based therapy
* Greater than or equal to 50% reduction in M-Protein sustained for a minimum of 60 days and no evidence of progression of disease while on the most recent course of VELCADE-based therapy
* 60 days or more since the patient's last VELCADE dose
* Life expectancy > 3 months
* Progressive disease defined by new or worsening lytic bone lesions or plasmacytoma or hypercalcemia or a >25% increase in M-protein

Exclusion Criteria:

* No patients with progressive disease while receiving an anthracycline-based regimen
* No patients with >2 prior regimens for the treatment of multiple myeloma
* No major surgery within 2 weeks before screening
* No patients with history of allergic reaction to compounds containing boron, mannitol, anthracycline, or liposomal formulations of any agent
* No patients known to be human immunodeficiency virus (HIV) positive
* No patients with poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness
* No patients with an active systemic infection requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the overall response rate defined as the partial or complete response to treatment according to EBMT criteria. Overall response will be assessed at each treatment cycle up to 8 cycles. | Assessed at each 21-day treatment cycle up to 8 cycles and over 6 months following discontinuation of all study drugs.

SECONDARY OUTCOMES:
Secondary endpoints include time to disease progression (treatment start to disease progression or death due to progression); best response assessed by the investigator; duration of response; and overall survival (treatment start to death by any cause). | Day 1, Cycle 1 throughout treatment cycles and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.